CLINICAL TRIAL: NCT00356811
Title: An Open-label, Single-arm, Multi-centre, Phase II Study of Oral Lapatinib in Combination With Paclitaxel as First-line Treatment for ErbB2-amplified Metastatic Breast Cancer Patients
Brief Title: Lapatinib Combined With Paclitaxel For Patients With First-Line ErbB2-Amplified Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF105764
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-05

CONDITIONS: Neoplasms, Breast
Keywords: Lapatinib; Metastatic breast cancer; Paclitaxel; ErbB2-amplification; GW572016
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Subjects will receive a daily dose of lapatinib until disease progression or withdrawal from study treatment due to unacceptable toxicity or withdrawal of consent. Subjects will be treated with paclitaxel for at least 6 months, and may continue on paclitaxel at the discretion of the Investigator, or discontinued sooner if the subject has disease progression, an unacceptable toxicity or withdraws consent.
  Interventions: Drug: Lapatinib oral tablets; Drug: Paclitaxel infusion

INTERVENTIONS:
Drug: Lapatinib oral tablets — Lapatinib will be given as tablets contain 410 mg of lapatinib ditosylate monohydrate, equivalent to 250 mg lapatinib free base per tablet. Subjects will be given a 4 week supply of lapatinib tables and instructed to take 6 tablets daily (1500 mg daily dose) orally at the same time each day. Subjects will receive a daily dose of lapatinib until disease progression or withdrawal from study treatment due to unacceptable toxicity or withdrawal of consent.
  Other Names: Tykerb/ Tyverb
Drug: Paclitaxel infusion — Subjects will receive weekly paclitaxel (80 mg/m2 IV for 3 weeks in a 4 week cycle). Subjects will be treated with paclitaxel for at least 6 months, and may continue on paclitaxel at the discretion of the Investigator, or discontinued sooner if the subject has disease progression, an unacceptable toxicity or withdraws consent.
  Other Names: Taxol

SUMMARY:
This study investigates the safety and efficacy of oral lapatinib in combination with an approved medication, paclitaxel, for patients with ErbB2 metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Signed informed consent.
* Only females ≥18 years of age will be recruited:

  * Non-child-bearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation or hysterectomy, or women who are postmenopausal); or
  * Child-bearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhoea (severe), women who are perimenopausal and young women who have begun to menstruate. These subjects must provide a negative serum pregnancy test at Screening and agree to one of the following:
  * Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication; or
  * Consistent and correct use of one of the following acceptable methods of birth control:
  * Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject.
  * Implants of levonorgestrel.
  * Injectable progestogen.
  * Any intrauterine device (IUD) with a documented failure rate of less than 1% per year.
  * Oral contraceptives (either combined or progestogen only).
  * Barrier methods, including diaphragm or condom with a spermicide.
* Subjects must have histologically confirmed invasive breast cancer with stage IVdisease;

  • Where the disease is restricted to a solitary lesion, the neoplastic nature of the lesion should be confirmed by cytology or histology.
* Subjects whose disease is ER+ and/or PR+ or unknown status will only be included in the study if they meet the following criteria:

  * They have symptomatic visceral disease that requires chemotherapy (e.g., patients with liver or lung metastases).
  * The disease is considered by the Investigator to be progressing rapidly or lifethreatening.
  * Subjects who have received endocrine therapy and who are no longer benefiting from this therapy.
* Documented amplification of ErbB2 defined by FISH in primary or metastatic tumor tissue. Results of FISH testing at local laboratories are acceptable, however, tissue sample must still be sent to Central laboratory where results will be repeated but not used for eligibility criterion.
* If a taxane had been administered in the neoadjuvant or adjuvant setting, progression must have occurred ≥12 months after completion of this treatment.
* Measurable lesion(s) according to RECIST (Response Evaluation Criteria in Solid Tumors) criteria [Stephens, 2004; Therasse, 2000].
* Radiotherapy prior to initiation of study medication is allowed to a limited area (e.g., palliative treatment for painful bone metastases), if it is not the sole site of disease. Subject must have completed radiation treatment and recovered from all acute radiation treatment-related toxicities, in particular bone marrow suppression.
* Bisphosphonate therapy for bone metastases is allowed however; treatment must be initiated prior to the first dose of study medication. Prophylactic use of bisphosphonates in subjects without bone disease, except for the treatment of osteoporosis, is not permitted.
* Subjects with stable central nervous system (CNS) metastases (stable for at least 3 months) as confirmed by computerized tomography (CT)/magnetic resonance imaging (MRI)) or leptomeningeal involvement are eligible only if they are not taking oral steroids or enzyme-inducing anticonvulsants.
* Subjects must have a cardiac ejection fraction within institutional range of normal as measured by echocardiogram (or multigated acquisition (MUGA) scan if an echocardiogram cannot be performed or is inconclusive). Subjects with known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure are not eligible.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 1.
* Considered by the Investigator to have a life expectancy of at least 3 months.
* Able to swallow and retain oral medication.
* Subjects must have new or archived tumor tissue available for analysis.
* Subjects must complete all screening assessments as outlined in the protocol.
* Subject must have adequate organ function as defined in Table 1.

Table 1 Baseline Laboratory Values for Adequate Organ Function SYSTEM LABORATORY VALUES

Haematologic

Absolute neutrophil count ≥1.5 × 10^9/L Haemoglobin ≥9 g/dL Platelets ≥100 × 10^9/L

Hepatic

Albumin ≥2.5 g/dL Serum bilirubin

* 1.25 x ULN AST and ALT ≤3 × ULN without liver metastases
* 5 × ULN with documented liver metastases

Renal

Serum Creatinine1 ≤2.0 mg/dL

* OR - Calculate Creatinine Clearance1 ≥40 mL/min

  1. Calculated by the Cockcroft and Gault Method. ALT = alanine aminotransferase; AST = aspartate aminotransferase

     Exclusion Criteria:

     A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Pregnant or lactating females.
* Received prior chemotherapy, hormonal therapy, immunotherapy, biologic therapy for metastatic disease.
* Prior therapy with ErbB1 and/or ErbB2 inhibitors.
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy) while taking study medication.
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment.
* Peripheral neuropathy of grade 2 or greater.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded.
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety.
* Active or uncontrolled infection.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure.
* Concurrent treatment with an investigational agent or participation in another clinical trial involving investigational agents.
* Used an investigational drug within 30 days or five half-lives, whichever is longer, preceding the first dose of investigational treatment.
* The subject has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to lapatinib or excipients and those related to paclitaxel or excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Latvia (2):
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Riga
- Poland (3):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, Bucharest, Romania
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg

REFERENCES:
- [Background] Jagiello-Gruszfeld A, Tjulandin Sergei S, Dobrovolskaya N et al, Lapatinib (L) with weekly paclitaxel (P) as first-line therapy for patients (pts) with HER2+ metastatic breast cancer (MBC). The 31st Annual San Antonio Breast Cancer Symposium; San Antonio TX: December 10-14 2008. Abstract 3145.
- [Background] Jagiello-Gruszfeld A, Tjulandin S, Dobrovolskaya N, Manikhas A, Pienkowski T, DeSilvio M, Ridderheim M, Abbey R. A single-arm phase II trial of first-line paclitaxel in combination with lapatinib in HER2-overexpressing metastatic breast cancer. Oncology. 2010;79(1-2):129-35. doi: 10.1159/000318043. Epub 2010 Nov 22. PMID 21088439

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib With Paclitaxel: Participants received lapatinib 1500 milligrams (mg) orally once daily (OD) with paclitaxel, administered as a 1-hour intravenous (IV) infusion at a dose of 80 mg/meters squared (m^2) on Days 1, 8, and 15 (±2 days) of a 28-day treatment cycle for at least 6 months. Participants were treated until disease progression, unacceptable toxicity, or consent withdrawal.
Period: Overall Study
Arm/Group | Lapatinib With Paclitaxel
Started | 57
Completed | 8
Not Completed | 49
Not completed — Death | 35
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 6
Not completed — Participant Could Not Make a Checkup | 1
Not completed — Study Is Terminating | 3
Not completed — Site Closed during Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Lapatinib Plus Paclitaxel: Participants received lapatinib 1500 mg orally OD with paclitaxel, administered as a 1-hour IV infusion at a dose of 80 mg/m^2 on Days 1, 8, and 15 (±2 days) of a 28-day treatment cycle for at least 6 months. Participants were treated until disease progression, unacceptable toxicity, or consent withdrawal.
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Best Overall Response (OR) of Confirmed Complete Response (CR) or Partial Response (PR), as Assessed by the Independent Review Committee (IRC)
Description: OR is defined as the number of participants achieving either a CR or PR, per Response Evaulation Criteria in Solid Tumors (RECIST). The best OR is defined as the best response recorded from the start of treatment until progressive disease (PD)/recurrence. CR is defined as the disappearance of all target lesions (TLs) and non-TLs. PR is defined as at least a 30% decrease in the sum of the longest diameters (LD) of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of one or more non-TL(s), as assessed by the IRC. PD is defined as at least a 20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs. Responses were confirmed at subsequent assessments made >=28 days after the original response. Participants with an unknown or missing response are treated as non-responders.
Time Frame: From the first dose of study medication to the first documented evidence of a confirmed CR or PR (up to Week 86)
Population: Intent-to-Treat (ITT) Population: all participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 57
Participants
  CR | 0
  PR | 29
Statistical Analysis 1: Comparison: Lapatinib Plus Paclitaxel; Test type: Superiority or Other; percentage of participants = 50.9, 95% CI 2-sided [37.3 to 64.4] — The estimated value represents the percentage of participants with a confirmed CR or PR

2. Secondary Outcome: Number of Participants With a Best Overall Response (OR) of Confirmed Complete Response (CR) or Partial Response (PR), as Assessed by the Investigator
Description: OR is defined as the number of participants achieving either a CR or PR, per RECIST. The best OR is defined as the best response recorded from the start of treatment until progressive disease (PD)/recurrence. CR is defined as the disappearance of all target lesions (TLs) and non-TLs. PR is defined as at least a 30% decrease in the sum of the longest diameters (LD) of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of one or more non-TL(s), as assessed by the Investigator. PD is defined as at least a 20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs. Responses were confirmed at subsequent assessments made >=28 days after the original response. Participants with an unknown or missing response are treated as non-responders.
Time Frame: From the first dose of study medication to the first documented evidence of a confirmed CR or PR (up to Week 86)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 57
Participants
  CR | 3
  PR | 41

3. Secondary Outcome: Duration of Response (DoR), as Assessed by the IRC
Description: DoR is defined for the subset of participants who had a confirmed CR (disappearance of all TLs and non-TLs) or PR (>=30% decrease in the sum of the LD of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of one or more non-TL[s]) as the time from the first documented evidence of a CR or PR until the first documentation of radiological PD or death due to breast cancer, if sooner. PD is defined as a >=20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs. For participants who did not progress or die, DoR was censored on the date of the last radiological scan. If a participant had only a Baseline visit or did not have a date of a radiological scan that was later than the date of initiation of anti-cancer therapy, DoR was censored at the start date of treatment.
Time Frame: From the first documented evidence of a PR or CR until the earlier of the date of disease progression or the date of death due to breast cancer (up to Week 86)
Population: ITT Population. Only those participants with CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Overall Study Arm: Participants received lapatinib 1500 mg orally OD with paclitaxel, administered as a 1-hour IV infusion at a dose of 80 mg/m^2 on Days 1, 8, and 15 (±2 days) of a 28-day treatment cycle for at least 6 months. Participants were treated until disease progression, unacceptable toxicity, or consent withdrawal.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 29
weeks | 39.7 [26.9 to 50.0]

4. Secondary Outcome: Duration of Response (DoR), as Assessed by the Investigator
Description: as for outcome 3
Time Frame: as for outcome 3
Population: ITT Population. Only those participants with CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 44
Weeks | 42.3 [37.7 to 64.1]

5. Secondary Outcome: Time to Response, as Assessed by the IRC
Description: Time to response is defined as the time from randomization until the first documented evidence of a PR or CR (whichever status is recorded first). Analysis was based on responses confirmed at a repeat assessment made at least 4 weeks after the initial response, with the time to response taken as the first time the response was observed, not the confirmation assessment. Participants who withdraw with no tumor response were censored at the date of withdrawal from the study. CR is defined as the disappearance of all TLs and non-TLs. PR is defined as at least a 30% decrease in the sum of the LD of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of one or more non-TL(s). PD is defined as at least a 20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs.
Time Frame: From randomization until the first documented evidence of a PR or CR (up to Week 86)
Population: ITT Population. Only those participants with CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 29
weeks | 8.4 [7.9 to 11.1]

6. Secondary Outcome: Time to Response, as Assessed by the Investigator
Description: as for outcome 5
Time Frame: From randomization until the first documented evidence of a PR or CR (up to Week 86)
Population: ITT Population. Only those participants with CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 44
Weeks | 8.0 [7.9 to 8.1]

7. Secondary Outcome: Time to Progression, as Assessed by the IRC and the Investigator
Description: Time to progression is defined as the interval between the start date of treatment and the date of radiological disease progression or death due to breast cancer, whichever occurs first. Participents who did not progress or die were censored on the date of their last radiological assessment preceding the start of any additional anti-cancer therapy. PD is defined as at least a 20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs. Responses were confirmed at a subsequent assessment made no less than 28 days after the original response.
Time Frame: From the start date of treatment until the date of radiological disease progression or the date of death due to breast cancer (up to Week 86)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 57
weeks
  IRC | 47.9 [40.0 to NA] — The upper limit of the 95% confidence interval could not be determined (not reached) because there were not enough events to be able to calculate it.
  Investigator | 50.9 [47.0 to 64.3]

8. Secondary Outcome: Progression-free Survival, as Assessed by the IRC and the Investigator
Description: Progression-free survival is defined as the interval between the start date of treatment and the date of radiological disease progression or death due to any cause, whichever occurs first. Participants who did not progress in their disease were censored on the date of their last radiological assessment preceding the start of any additional anti-cancer therapy. PD is defined as at least a 20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs. Responses were confirmed at a subsequent assessment made no less than 28 days after the original response.
Time Frame: From the start date of treatment until the date of radiological disease progression or death due to any cause, whichever occurs first (up to Week 86)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 57
weeks
  IRC | 47.9 [40.0 to NA] — The upper limit of the 95% confidence interval could not be determined (not reached) because there were not enough events to be able to calculate it.
  Investigator | 50.9 [47.0 to 64.3]

9. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the interval between the date of treatment start and the date of death due to any cause. For participants who did not die, follow-up was censored as the date of last contact. For participants who did not die, follow-up was censored at the date of last contact.
Time Frame: From the date of the first dose until the date of death due to any cause (up to Week 86)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 57
weeks | NA [NA to NA] — At the time of this analysis, the median and the 95% confidence interval could not be determined because there were not enough deaths to calculate these estimates.

10. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment was exercised in deciding whether reporting was appropriate in other situations.
Time Frame: From the start of study medication until 28 days after the last dose (up to Study Week 381)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Lapatinib Plus Paclitaxel
Number analyzed (Participants) | 57
Participants
  Any AE | 57
  Any SAE | 11

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until 28 days after the last dose (up to Study Week 381).
Description: SAEs and non-serious AEs are reported for members of the ITT Population, comprised of all participants who received study medication.
Arm/Group | Lapatinib Plus Paclitaxel
Serious Adverse Events (participants affected / at risk) | 11/57
Other Adverse Events (participants affected / at risk) | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Paclitaxel (N=57)
Neutropenia (Blood and lymphatic system disorders) | 4
Abscess limb (Infections and infestations) | 1
Abscess soft tissue (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Cardiopulmonary failure (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Paclitaxel (N=57)
Diarrhoea (Gastrointestinal disorders) | 32
Neutropenia (Blood and lymphatic system disorders) | 25
Rash (Skin and subcutaneous tissue disorders) | 23
Fatigue (General disorders) | 15
Peripheral sensory neuropathy (Nervous system disorders) | 14
Leukopenia (Blood and lymphatic system disorders) | 10
Alanine aminotransferase increased (Investigations) | 10
Anaemia (Blood and lymphatic system disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 9
Neuropathy peripheral (Nervous system disorders) | 8
Vomiting (Gastrointestinal disorders) | 6
Oedema peripheral (General disorders) | 6
Upper respiratory tract infection (Infections and infestations) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 6
Asthenia (General disorders) | 5
Erysipelas (Infections and infestations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Hypersensitivity (Immune system disorders) | 4
Weight decreased (Investigations) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Paronychia (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 3
Headache (Nervous system disorders) | 3
Nail dystrophy (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.